CLINICAL TRIAL: NCT07288684
Title: Chiropractor Delivered Virtual Intervention After Vertebral frActure (VIVA)
Brief Title: Chiropractor Delivered Virtual Intervention After Vertebral frActure
Acronym: VIVA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Waterloo (Other)
Collaborators: Canadian Chiropractic Research Foundation (Unknown); Canadian Chiropractic Association, Canadian Chiropractic Research Foundation (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Health Services Research
Other Study IDs: CTO 4816
Record Dates: First submitted 2025-07-16; First posted 2025-12-17 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-10

CONDITIONS: Osteoporosis; Vertebral Fracture
Keywords: Rehabilitation
MeSH Terms: conditions — Osteoporosis; Spinal Fractures

STUDY DESIGN:
Intervention Model Description: We will conduct a pragmatic, pilot trial with two parallel groups with a 1:1 ratio.
  Participants will be randomized to: 1) immediate receipt of VIVA intervention; or 2) waitlist usual care control and delayed receipt of VIVA 10 weeks post-randomization.
Who Masked: Outcomes Assessor
Masking Description: Outcome assessors will be blind to group allocation. Participants will not be blind to group allocation because they will know what group they are assigned to.
  The waitlist control was chosen based on input from persons with lived experience, who indicated that participants may be more willing to participate if there was a wait list control rather than receiving no intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Immediate Receipt of VIVA (Experimental): Participants receive a technology consultation 1-2 weeks prior to baseline assessment, and receive intervention in week one (immediately post-randomization).
  Following a virtual assessment, participants will receive twelve 1:1 virtual sessions (via Zoom) over eight weeks.
  Interventions: Behavioral: VIVA
- Control (No Intervention): Participants receive a technology consultation 1-2 weeks prior to baseline assessment, and receive intervention in week ten (waitlist control).

INTERVENTIONS:
Behavioral: VIVA — VIVA is an intervention for people with vertebral fractures that covers four areas: pain management, safe movement, exercise, and nutrition. It includes print and video resources, and a framework for goal setting, selecting exercises, and teaching body mechanics.
  Arms: Immediate Receipt of VIVA

SUMMARY:
This study will determine feasibility of a chiropractor delivered virtual intervention for individuals following osteoporotic vertebral fracture.

This pilot trial will have two parallel groups with a 1:1 ratio. Participants will be randomized to: 1) immediate receipt; or 2) waitlist usual care control and delayed receipt of VIVA 10 weeks post-randomization.

VIVA is an intervention for people with vertebral fractures that covers four areas: pain management, safe movement, exercise, and nutrition. It includes print and video resources, and a framework for goal setting, selecting exercises, and teaching body mechanics.

A chiropractor (DC) completes a virtual assessment and then leads twelve 1:1 virtual sessions (via Zoom) over eight weeks. Sessions start with brief education on a topic (e.g., safe movement, pain management, exercise, nutrition), followed by training and modeling of exercise and safe movement strategies, then goal setting, and action planning.

This trial will be considered feasible if a) we recruit 14 people in eight months; b) 80% of participants complete the trial; and c) exercise adherence is 75%.

DETAILED DESCRIPTION:
Spine fractures are the most common fracture due to osteoporosis. They can happen because of falls or activities of daily life like bending and lifting. Fractures of the spine can result in pain, which can last for a long time. Spine fractures can affect breathing, appetite, digestion, and mobility, and can restrict or modify an individuals' work or daily activities.

There are no standard rehabilitation programs after spine fracture, and patients often must pay out of pocket for rehabilitation. Rehabilitation can be hard to access (especially in rural or remote locations) and it can be difficult to find providers with training and expertise to treat spine fractures.

Our team includes Osteoporosis Canada, patients, health care professionals, and researchers from multiple provinces. We reviewed research, consulted patients and healthcare providers to understand their experiences with spine fracture rehabilitation to develop a Toolkit for a virtual rehabilitation program for people with spine fracture, called VIVA.

VIVA is an intervention for people with vertebral fractures that covers four areas: pain management, safe movement, exercise, and nutrition. It includes print and video resources, and a framework for goal setting, selecting exercises, and teaching body mechanics. We used the Behavior Change Wheel method to select four implementation strategies: education on pain management, safe movement, exercise, and nutrition; modeling of and training on exercises, safe movement, and pain management strategies; and enablement, such as goal setting, action planning, and self-monitoring.

Participants receive a technology consultation 1-2 weeks prior to baseline assessment, and receive intervention in week one (immediately post-randomization) or in week ten (waitlist control). A provider completes a virtual assessment, and then leads 1:1 once-weekly virtual sessions (via Zoom) over eight weeks. Sessions start with brief education on a topic (e.g., safe movement, pain management, exercise, nutrition), followed by training and modeling of exercise and safe movement strategies, then goal setting, and action planning.

The provider prescribes resources (e.g., summaries, pictures, videos) using the Wibbi app (https://wibbi.com/) or that can be emailed or mailed. Exercises are tailored to the participant's abilities, and target balance, muscle strength, and endurance of back extensor muscles and scapular stabilizers. The first session will serve as an intake session.

Depending on the patient needs the provider either will provide training on exercises, movement tips, or pain management tips. Finally, the provider will show how to monitor performance and adherence throughout the intervention, discuss and decide on the area of focus for the next session (i.e., pain management, safe movement, exercise, nutrition), and schedule the next session.

The remaining 11 sessions from Week 2 to Week 8 will start with education on the chosen topic. The provider will review progress on exercises, movement strategies, or pain management tips from the previous sessions and demonstrate new exercises or strategies. The provider will deliver the exercises prescribed and any educational resources through the Wibbi app and decide on an area of focus for the next session based on discussion with the participant.

VIVA was designed and user tested in the context of physiotherapist delivery, but chiropractors may be well-situated to deliver VIVA. Chiropractors and physiotherapists manage similar patient bases with overlapping scopes of practice. We propose a pilot study of the feasibility of the implementation of the VIVA Toolkit with a chiropractor as the provider (i.e., Can we recruit people? Do they like the program? Do they attend?). Through this study we will also collect information about pain, quality of life and physical functioning before and after the intervention. We will then use the findings of this study to determine if it is feasible to include chiropractor providers in a larger clinical trial.

ELIGIBILITY:
Inclusion Criteria:

* Over the age of 50 (men or post-menopausal women)
* Have had a vertebral fracture in the past two years
* Willing to participate in twelve (12) virtual rehabilitation sessions for 10 weeks
* Have access to internet and a smart device with a camera and microphone

Exclusion Criteria:

* Cauda equina syndrome or spinal cord injury
* Had a traumatic fracture (i.e., car accident)
* An active infection
* Active inflammatory arthritis with a flare up within the past two years
* An inability to follow two-step commands or understand instructions and are without a caregiver to support participation
* Been participating in a similar rehabilitation program for vertebral fractures delivered by a physical therapist, exercise physiologist or kinesiologist and includes exercise
* Any surgeries planned or health problems that might cause their health to change significantly in the next 3 months

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2025-10-20 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Feasibility of Chiropractic Delivery | We will consider ≥80% retention at 20 weeks acceptable. Adherence will be defined as ≥2 sessions per week of exercise at 20 weeks
  This trial will be considered feasible if a) we recruit 14 people in eight months; b) 80% of participants complete the trial; and c) exercise adherence is 75%.

SECONDARY OUTCOMES:
Participant experience | At completion of 10 weeks.
  We will lead exit interviews using an interview guide with open-ended questions guided by user-centred design principles.
Pain and Quality of Life | Will be measured at weeks 10/20 (effectiveness) and 20 weeks (sustainability, immediate group only
  Using the QUALEFFO-41 to measure health-related quality of life, the QUALEFFO-41 also includes questions on pain.
Health-Related Quality of life | Will be measured at weeks 10/20 (effectiveness) and 20 weeks (sustainability, immediate group only
  We will use the EuroQOL instrument (EQ5D5L) to measure health-related quality of life
Physical Performance - Balance | Physical performance will be measured at weeks 10/20 (effectiveness) and 20 (sustainability, immediate group only).
  We will assess static balance via three point balance scale from the Short Physical Performance Battery.
  Scoring:
  A. Side-by-side-stand Held for 10 sec ❒ 1 point Not held for 10 sec ❒ 0 points Not attempted ❒ 0 points
  Number of seconds held if less than 10 sec: _______ sec *If 0 points, end Balance Tests
  B. Semi-Tandem Stand Held for 10 sec ❒ 1 point Not held for 10 sec ❒ 0 points Not attempted ❒ 0 points
  Number of seconds held if less than 10 sec: _______ sec *If 0 points, end Balance Tests
  C. Tandem Stand Held for 10 sec ❒ 2 points Held for 3 to 9.99 sec ❒ 1 point Held for < than 3 sec ❒ 0 points Not attempted ❒ 0 points (circle reason above)
Physical Performance - Sit to Stand Performance | Physical performance will be measured at weeks 10/20 (effectiveness) and 20 (sustainability, immediate group only)
  We will assess sit-to-stand performance (30 Second Chair Stand Test).
  Test Instructions With your shoes on, complete as many repetitions as you can safely and at your own pace.
  Single Chair Stand (Practice)
  1. Sit in the middle of the chair.
  2. Keep your feet flat on the floor, hip width apart.
  3. Keep your back straight and hold your arms across the chest.
  4. Rise to a full standing position, then sit back down again.
  5. If you are able to complete one repetition safely, proceed with the full test on the next page. If not, this is the end of the test.
  Scoring: 30s Chair Stand Test AGE Men Women 60-64 < 14 < 12 65-69 < 12 < 11 70-74 < 12 < 10 75-79 < 11 < 10 80-84 < 10 < 9 85-89 < 8 < 8 90-94 < 7. < 4
Adherence to diet recommendations | Measured at 20 weeks, immediate group only
  Protein, calcium, vitamin D and energy intake will be measured with ASA24 and compared to Health Canada recommended dietary allowances.
Adverse events | On-going, disclosed during intervention sessions, or at assessment milestones (week 10 and 20).
  We will ask participants to report adverse events, defined using Health Canada definitions and established protocols. We will report all serious and non-serious adverse events (including falls, fractures) and identify them as: a) Expected/Unexpected and b) Related/unrelated to the intervention program.
  Participants instructed to inform chiropractor if they have an adverse event. "If you have an illness, injury, or need to get medical help, whether it is due to study participation or not, please contact us." During the week 10 and week 20 assessments, assessors to inquire about whether the participant had any illnesses or injuries.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Waterloo, Waterloo, Ontario, Canada